CLINICAL TRIAL: NCT03820544
Title: Preoperative Endoscopic Biliary Drainage With Self Expanding Metal Stents (SEMS) vs. Direct Surgical Resection for Patients With Severe Obstructive Jaundice
Brief Title: SEMS Placement Before Surgery in Unblocking Bile Duct in Patients With Periampullary Pancreatic Cancer With Severe Obstructive Jaundice
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interest in this study changed and it was decided to end enrollment early
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16D.759; JT 10199 (Other: JeffTrial Number)
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Results first posted 2019-10-10 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEMS (Experimental): Patients undergo Endoscopic Retrograde Cholangiopancreatography (ERCP) with Self Expanding Metal Stents (SEMS) placement before standard of care surgical resection.
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreatography
- Standard of care surgical resection (Active Comparator): Patients undergo standard of care surgical resection.
  Interventions: Other: Standard of care

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangiopancreatography — Undergo ERCP with SEMS placement
  Other Names: ERCP
  Arms: SEMS
Other: Standard of care — Undergo standard of care surgical resection
  Arms: Standard of care surgical resection

SUMMARY:
This trial studies the side effects of self expanding metal stent (SEMS) placement before surgery in unblocking the bile duct in patients with periampullary pancreatic cancer with severe obstructive jaundice. SEMS placement unblocks the bile duct and may help in improving bile drainage prior to surgery in patients with periampullary pancreatic cancer with severe obstructive jaundice.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the 30-day overall complication rates between patients with severe obstructive jaundice undergoing preoperative endoscopic biliary drainage with self expanding metal stents (SEMS) and patients undergoing direct surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of operable peri-ampullary pancreatic cancer as determined by the Department of Surgery per their standard of care
* Serum bilirubin > 10 mg/dl
* Adequate birth control

Exclusion Criteria:

* Patients with evidence of distant metastasis on computed tomography (CT) or magnetic resonance imaging (MRI)
* Patients anticipated to require vascular reconstruction
* Patients with cholangitis
* Patients for whom surgery is deemed inappropriate by surgeon
* Patients with bilirubin less than 10 mg/dL or greater than 20 mg/dL
* Patients who previously underwent biliary decompression for cholangitis by ERCP or percutaneous transhepatic cholangiography (PTC)
* Patients with low performance score (Karnofsky performance status scale < 50)
* Patients with known preexisting liver disease with associated elevated bilirubin
* Patients who are pregnant or actively breast feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kowalski, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SEMS | Standard of Care Surgical Resection
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SEMS | Standard of Care Surgical Resection | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Complication Rates of Grade III or Higher
Description: The risk difference will be calculated (stent minus control) with a one-sided 95% confidence interval.
Time Frame: At 30 days post-surgery
Population: Due to the low enrollment number to this study, statistical analysis was not conducted due to insufficient data collected to run analyses.
Arm/Group | SEMS | Standard of Care Surgical Resection
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Intraoperative Estimated Blood Loss
Description: Group comparisons will be performed using two sample t-tests or Wilcoxon rank sum tests.
Time Frame: At time of surgery
Population: as for outcome 1
Arm/Group | SEMS | Standard of Care Surgical Resection
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year after surgery
Arm/Group | SEMS | Standard of Care Surgical Resection
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03820544/Prot_SAP_000.pdf